CLINICAL TRIAL: NCT01153789
Title: Evaluation and Medical Care of Oculomotor Dysfunction Leading to Vertigo in Children
Brief Title: Study of Oculomotor Dysfunction Leading to Children Vertigo
Acronym: VERVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P081114
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2013-08

CONDITIONS: Vertigo; Headache; Anomaly of Vergence System; Accommodation Disorders; Orthoptic Rehabilitation
Keywords: Vergence-accommodation evaluation; Vergence and postural control; Dynamic visual acuity
MeSH Terms: conditions — Vertigo; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients orthoptic rehabilitation (Experimental): Children with vertigo-headache and vergence disorders
  Interventions: Procedure: orthoptic rehabilitation
- Control Orthoptic diagnostic (Other): Healthy controls
  Interventions: Other: Orthoptic diagnostic

INTERVENTIONS:
Procedure: orthoptic rehabilitation — Orthoptic rehabilitation: 12 sessions (2 sessions per week) At the end of a series of 12 sessions of orthoptic, the child will be examined and will again perform an static and dynamic oculomotor evaluation and control of postural balance.
  Arms: Patients orthoptic rehabilitation
Other: Orthoptic diagnostic — postural, oculomotor and orthoptics tests
  Arms: Control Orthoptic diagnostic

SUMMARY:
The eye movements of vergence allow binocular vision whatever the viewing distance or the body movements are and the perception of depth. Vergence dysfunction can lead to erroneous visual sensation of movements. In our daily life using screens (computer, game boys..) is increasing and this approach heavily the ocular vergence and can lead to symptoms if oculomotor and accommodative systems are dysfunctioning (Ped. Neurology 2000). Not knowing this pathology lead to inappropriate and expensive prescription CT scan or NMR. To evaluate the vergence performances just evaluation in static condition is currently available in ophthalmology departments. The CNRS laboratory (IRIS, FRE 3154) adapted a technic of eye movement recording to study ocular vergence in dynamic condition.

DETAILED DESCRIPTION:
The goals of the study are:

1. to compare the coordination of binocular eye movements, postural stability on a force-plate during visual tasks (looking at a target or reading) and dynamic visual acuity between two groups of children and teenagers: one group with oculomotor vergence disorders and vertigo and one group with normal eye movements. Children will undergo complete vestibular testing (by Dr WIENER-VACHER) to eliminate a vestibular origin for vertigo. Normal children will be volunteers.
2. in order to evaluate objectively the effect of rehabilitation, a second oculomotor evaluation (identical to the initial one) will be done in children with vertigo after an orthoptic rehabilitation focused on ocular vergence. We hypothesize that functional oculomotor disorders can be rehabilitated because of the plasticity of the oculomotor system (proved by several studies for many years) provided that the spatial temporal parameters of the training are precisely tailored to patient malfunction.
3. Establish normative data of the binocular eye movements and posturography, and validate a protocol for complete static and dynamic oculomotor evaluation for clinical use. To a longer term modification of the rehabilitation protocols of eye movements will be designed to fit each patient problems in function of the abnormalities revealed by the static and dynamic evaluation.

Study calendar :

All the children referred for vertigo with vergence abnormalities and normal vestibular functional evaluation will be proposed for participate to the study.

The patients included in the study will perform an oculomotor complete evaluation (static and dynamic and accommodation), posturography test and a visual dynamic acuity test. These tests will last for 60 minutes, including breaks to avoid fatigue of the children. Then, the children will follow orthoptic rehabilitation :12 sessions (2 sessions per week). These sessions will be done by an orthoptist installed close to home, in contact with the research team.

At the end of a series of 12 sessions of orthoptic, the child will be examined and will again perform a static and dynamic oculomotor evaluation and control of postural balance.

In order to highlight the prolonged effects of rehabilitation a third oculomotor evaluation and control of postural balance will be made six months after inclusion.

Healthy children (control group) will be recruited at Robert Debré hospital. A poster campaign in the corridors of the hospital, as well as general information (mailing) for the Hospital staff will be made.

A questionnaire prior to a half-hour will confirm the normal vestibular children. After completing the questionnaire, a test Postural oculomotor (one hour) and a test orthoptics (half hour) will be made.

Conduct of Research: We will study with a multidisciplinary approach children with vergence abnormalities and vertigo and/or headache. Healthy children will also be examined for baseline data.

Methodology :

Statistical analysis will be conducted at the Unite de Recherche Clinique Paris Nord, Robert Debré Hospital.

The qualitative data will be described in terms of frequency and percentages, quantitative data as mean (SD) if the distribution follows a normal distribution, as median (quartiles) otherwise. The influence of sex adjusted for age will be tested by parametric methods after normalization of distributions.

The establishment of standards will be conducted according to the method described by EM Wright et P. ROYSTON (Simplified estimation of age-specific reference intervals for skewed data, Statistics in Medicine 1997, vol 16, 2785-2803). The method is to produce smoothed percentile curves by time (age) using parametric methods.

Analysis of sick children will be purely descriptive. She will describe the differences for different standard deviation scores of variables described in the previous paragraph between the time of diagnosis and after 12 weeks of rehabilitation and orthoptic vergence.

ELIGIBILITY:
Inclusion Criteria:

* Children with disorders of vergence:

  * 6 to 17 years old
  * Patient receiving a social security scheme
  * Presenting vergence problems (diagnosed by standard methods : prism bar using the proximal point of convergence and phoria) and suffering from vertigo and/or headache
  * Presenting anormal refraction
  * Free from any type vestibular pathology, ENT or neurological
  * Free from strabismus
  * Child and holders of parental authority have signed a consent

Healthy Children :

* 6 to 17 years old
* Free from any type of vestibular pathology, ENT or neurological
* Free from any type of neuron-ophthalmic/orthoptic pathology
* Child and holders of parental authority have signed a consent

Exclusion Criteria:

* Patient with a disease which (from the assessment of the investigator) could disrupt the monitoring or be disrupted by the participation in the study,

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 183 (Actual)
Dates: Start 2010-09; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
oculomotor complete evaluation (static and dynamic and accommodation), posturography test and a visual dynamic acuity test | t=0, t=3months, t=6months

SECONDARY OUTCOMES:
free of symptoms | t=3months, t=6months

CONTACTS AND LOCATIONS:
Overall Officials: Sylvette R WIENER, M.D., PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Thierry VAN DEN ABBEELE, M.D., PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- ORL Service - Robert Debre Hospital, Paris, Paris, France